CLINICAL TRIAL: NCT03561012
Title: Use of Team-Based Goals and Incentives to Improve the Performance of Community-Based Health Workers in Promoting Reproductive, Maternal, Newborn and Child Health and Nutrition Behaviors in Bihar, India: A Cluster Randomized Trial
Brief Title: Team-Based Goals and Incentives for Community-Based Health Workers to Promote Maternal and Child Health in Bihar, India
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Gary Darmstadt, Associate Dean for Maternal and Child Health, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: TBGI
Record Dates: First submitted 2018-06-06; First posted 2018-06-19 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Healthy
Keywords: health; nutrition; pregnancy; infant; child

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental)
  Interventions: Behavioral: Team-Based Goals and Incentives
- Control Arm (Active Comparator)
  Interventions: Other: Control Condition

INTERVENTIONS:
Behavioral: Team-Based Goals and Incentives — The intervention included 3 main components. 1) The intervention fostered a sense of team collective responsibility and solidarity (TEAM) by emphasizing the value of teamwork and front-line community health workers (FLWs) reciting a pledge at meetings to serve beneficiaries. 2) To establish goals and coverage targets related to maternal and child health outcomes (GOALs), 7 targets were identified related to delivery preparations, newborn care, exclusive breastfeeding, and family planning. 3) Small non-cash incentives were awarded to FLWs each quarter if their team met greater than 70% of the collective subcenter goals; incentives were most common cookware products (e.g., dish, cooking vessel, steamer). Non-cash incentives also included a certificate of recognition for teams that met their targets in all quarters (INCENTIVES). In the areas of the intervention and control arms, the Ananya program was also underway (see Brief Summary of the project).
  Arms: Intervention arm
Other: Control Condition — Standard of care
  Arms: Control Arm

SUMMARY:
This study is designed to evaluate the impact of team-based goals and performance-based incentives for community-based health workers on health-promoting behaviors among women related to reproductive, maternal, newborn and child health and nutrition in Bihar, India.

The intervention was funded by the Bill and Melinda Gates Foundation (BMGF) and implemented from 2012 to 2014. Health sub-centers in the catchment areas of five blocks (sub-districts) of the district of Bengusarai were randomly assigned to treatment or control arms (38 sub-centers were assigned to each). Data were collected in the Intervention and Control areas from mothers of infants 0-12 months at baseline and at 2.5-year follow-up, to assess the intervention's effects on quality and quantity of FLW home visits, postnatal health behaviors, and among older infants/toddlers, complementary feeding and vaccination. Difference in difference analyses were used to assess outcome effects in this quasi experimental study.

The TBGI intervention was implemented in areas where the BMGF-funded Ananya program (official title: Bihar Family Health Initiative) was also being implemented. Thus, the impact is of the [TBGI intervention + Ananya] versus [Ananya alone]. The Ananya program was developed and implemented via a partnership of BMGF and the Government of Bihar. The ultimate purpose of Ananya was to reduce maternal, newborn, and child mortality; fertility; and child undernutrition in Bihar, India. Ananya involved multi-level interventions designed to build front line health worker (FLW) capacities and reach to communities and households, as well as to strengthen public health facilities and quality of care to improve maternal and neonatal care and health behaviors, and thus survival. It was implemented from 2012 to 2014. Eight focal districts in western and central Bihar received Ananya, while 30 districts did not.

ELIGIBILITY:
Inclusion Criteria:

* Mothers of infants 0-12 months residing in the catchment area of the subcenters (public health facilities)

Exclusion Criteria:

-

Ages: 15 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3581 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2014-11-30 (Actual); Study Completion 2014-11-30 (Actual)

PRIMARY OUTCOMES:
At least 2 antenatal home visits in final trimester | Up to 2.5 years
  Assessed via self-report from representative sample of mothers of children aged 0-11 months.
At least one home visit within 24 hours of delivery, among women who had a home delivery | 2.5 year follow-up
  Assessed via self-report from representative sample of mothers of children aged 0-11 months.
At least one home visit within 1 week of delivery | 2.5 year follow-up
  Assessed via self-report from representative sample of mothers of children aged 0-11 months.
Complementary feeding home visit for women with infant 6-11 months old | 2.5 year follow-up
  Assessed via self-report from representative sample of mothers of children aged 0-11 months.
Postpartum family planning home visits | 2.5 year follow-up
  Assessed via self-report from representative sample of mothers of children aged 0-11 months.
Obtained phone number for delivery (Frontline worker's (FLW) number, number for private vehicle, number for ambulance, any of the above) | 2.5 year follow-up
  Assessed via self-report from representative sample of mothers of children aged 0-11 months.
Received 90 IFA tablets | 2.5 year follow-up
  Assessed via self-report from representative sample of mothers of children aged 0-11 months.
Immediate breastfeeding (within 1 hour of delivery) | 2.5 year follow-up
  Assessed via self-report from representative sample of mothers of children aged 0-11 months.
Nothing applied to the cord after cutting | 2.5 year follow-up
  Assessed via self-report from representative sample of mothers of children aged 0-11 months.
Infant age 6-11 months old ate cereal-based meal in previous day | 2.5 year follow-up
  Assessed via self-report from representative sample of mothers of children aged 6-11 months.
Current use of any modern method of contraception: | 2.5 year follow-up
  Assessed via self-report from representative sample of mothers of children aged 0-11 months.
Child age 6-11 months old received DPT3 vaccination | 2.5 year follow-up
  Assessed via self-report from representative sample of mothers of children aged 6-11 months.